CLINICAL TRIAL: NCT03564444
Title: A Phase 4, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Safety of 2 New of 6:2 Influenza Virus Reassortants in Adults
Brief Title: D2560C00015 FluMist Annual Safety Study 2018
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D2560C00015
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Influenza; Healthy
Keywords: Bivalent.; Influenza.; FluMist Quadrivalent.; Vaccine Prevention in Healthy Adults.
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bivalent influenza vaccine (Experimental): A single dose of bivalent vaccine (10^7±5 fluorescent focus unit of 2 cold-adapted, attenuated, temperature-sensitive, 6:2 reassortant influenza strain) will be administered as intranasal spray on Day 1
  Interventions: Biological: Bivalent influenza vaccine
- Placebo (Placebo Comparator): A single dose of placebo matched to bivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Bivalent influenza vaccine — A single dose of bivalent vaccine (10^7±5 fluorescent focus unit of 2 cold-adapted, attenuated, temperature-sensitive, 6:2 reassortant influenza strain) will be administered as intranasal spray on Day 1.
  Arms: Bivalent influenza vaccine
Other: Placebo — A single dose of placebo matched to bivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Arms: Placebo

SUMMARY:
This prospective annual release study is designed to evaluate the safety of 2 new influenza virus vaccine strains to be included in FluMist Quadrivalent for the 2018-2019 influenza season.

DETAILED DESCRIPTION:
This prospective. randomized, double-blind. placebo-controlled release study will enroll approximately 300 healthy adults 18 to 49 years of age (not yet reached their 50th birthday). Eligible subjects will be randomly assigned in a 4:1 fashion to receive a single dose of bivalent vaccine or placebo by intranasal spray. Randomization will be stratified by site. This study will be conducted at 2 sites in the United States of America. Each subject will receive 1 dose of investigational product on Day 1. The duration of study participation for each subject is the time from study vaccination through 180 days after study vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 49 years
* Written informed consent
* Subject available by telephone
* Ability to understand and comply with the requirements of the protocol, as judged by the Investigator

Exclusion Criteria:

* Concurrent enrollment in another clinical study up to 180 days after receipt of investigational product (Day 181)
* History of hypersensitivity to any component of the vaccine, including egg or egg protein or serious, life threatening, or severe reactions to previous influenza vaccinations
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (example (eg], asthma), chronic metabolic diseases (eg, diabetes mellitus), renaldysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (greater than [>]100.0 degrees Fahrenheit [F] oral or equivalent) and/or clinically significant respiratory illness (example, cough or sore throat) within 14 days to randomization
* Any known immunosuppressive condition or immune deficiency diseases, including human immunodeficiency virus infection, or ongoing immunosuppressive therapy
* History of Guillain-Barre syndrome.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Segall, MD, Principal Investigator — Clinical Research Atlanta; Keith Klatt, MD, Principal Investigator — Columbia Research Group
Locations (2):
- United States (2):
  - Research Site, Stockbridge, Georgia
  - Research Site, Portland, Oregon

REFERENCES:
- See also: Protocol and Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2560C00015&attachmentIdentifier=8e50bdf3-f051-45ee-a9e9-e40b1d25de6c&fileName=d2560c00015-csp-v1_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 06Jun2018 and 27Dec2018 in the USA.
Groups:
- Placebo: Participants received a single dose of placebo matched to bivalent vaccine by intranasal spray.
- Bivalent Vaccine: Participants received a single dose of bivalent vaccine by intranasal spray.
Period: Overall Study
Arm/Group | Placebo | Bivalent Vaccine
Started | 60 | 240
Completed | 60 | 240
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized and treated participants, grouped according to actual treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bivalent Vaccine | Total
Number analyzed (Participants) | 60 | 240 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.5 (8.6) | 30.5 (8.9) | 30.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 139 | 173
  Male | 26 | 101 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 12 | 16
  Not Hispanic or Latino | 56 | 228 | 284
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 12 | 52 | 64
  White | 47 | 167 | 214
  More than one race | 0 | 11 | 11
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Fever (Oral Temperature >= 101 Degrees Fahrenheit) Through Day 8
Description: Percentage of participants with fever (oral temperature >= 101 degrees Fahrenheit) through Day 8 is reported.
Time Frame: Day 1 through Day 8
Population: The ITT population included all randomized and treated participants, grouped according to actual treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Bivalent Vaccine
Number analyzed (Participants) | 60 | 240
Percentage of participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Bivalent Vaccine; Test type: Superiority; Risk Difference (RD) = 0, 95% CI 2-sided [-6.7 to 1.9]

2. Secondary Outcome: Number of Participants With Solicited Symptoms Through Day 8
Description: For this study, solicited symptoms included oral fever (> 100 degrees Fahrenheit), runny nose, sore throat, cough, vomiting, muscle aches, chills, decreased activity (tiredness), and headache.
Time Frame: Day 1 through Day 8
Population: The ITT population included all randomized and treated participants, grouped according to actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bivalent Vaccine
Number analyzed (Participants) | 60 | 240
Participants
  >100 degrees Fahrenheit | 0 | 0
  >102 degrees Fahrenheit | 0 | 0
  >103 degrees Fahrenheit | 0 | 0
  Runny nose | 4 | 33
  Sore throat | 2 | 14
  Cough | 3 | 7
  Vomiting | 1 | 0
  Muscle aches | 0 | 7
  Chills | 0 | 3
  Decreased activity (tiredness) | 2 | 9
  Headache | 6 | 27

3. Secondary Outcome: Number of Participants With Solicited Symptoms Through Day 15
Description: as for outcome 2
Time Frame: Day 1 through Day 15
Population: The ITT population included all randomized and treated participants, grouped according to actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bivalent Vaccine
Number analyzed (Participants) | 60 | 240
Participants
  >100 degrees Fahrenheit | 0 | 1
  >=101 degrees Fahrenheit | 0 | 1
  >102 degrees Fahrenheit | 0 | 1
  >103 degrees Fahrenheit | 0 | 0
  Runny nose | 4 | 37
  Sore throat | 4 | 17
  Cough | 3 | 9
  Vomiting | 1 | 0
  Muscle aches | 0 | 8
  Chills | 0 | 4
  Decreased activity (tiredness) | 3 | 13
  Headache | 8 | 33

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Through Day 8 and Day 15
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 8; Day 1 through Day 15
Population: The ITT population included all randomized and treated participants, grouped according to actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bivalent Vaccine
Number analyzed (Participants) | 60 | 240
Participants
  TEAEs through Day 8 | 1 | 15
  TEAEs through Day 15 | 2 | 19

5. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs) Through Day 29 and Day 181
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 29; Day 1 through Day 181
Population: The ITT population included all randomized and treated participants, grouped according to actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bivalent Vaccine
Number analyzed (Participants) | 60 | 240
Participants
  TESAEs through Day 29 | 0 | 1
  TESAEs through Day 181 | 0 | 1

6. Secondary Outcome: Number of Participants With New Onset Chronic Diseases (NOCDs) Through Day 29 and Day 181
Description: An NOCD is a newly diagnosed medical condition that is of a chronic, ongoing nature and is assessed by the investigator as medically significant.
Time Frame: Day 1 through Day 29; Day 1 through Day 181
Population: The ITT population included all randomized and treated participants, grouped according to actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bivalent Vaccine
Number analyzed (Participants) | 60 | 240
Participants
  NOCDs through Day 29 | 0 | 0
  NOCDs through Day 181 | 0 | 0

ADVERSE EVENTS:
Time Frame: For SAEs: Day 1 through Day 181 For non-serious AEs: Day 1 through Day 15
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience(immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Arm/Group | Placebo | Bivalent Vaccine
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/240
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/240
Other Adverse Events (participants affected / at risk) | 2/60 | 19/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Bivalent Vaccine (N=240)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Bivalent Vaccine (N=240)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT03564444/Prot_SAP_000.pdf